CLINICAL TRIAL: NCT00273767
Title: Double-blind Phase II Pilot Monocentric Randomized Clinical Trial Evaluating the Effect of a Preliminary Administration of Erythropoietin on Different Markers of Cardiac Ischemia Induced by Cardiopulmonary Bypass
Brief Title: Preliminary Administration of EPO and Markers of Cardiac Ischemia Induced by CPB
Acronym: EPOetCEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Frédérick Marie, University Hospital Grenoble
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DCIC 05 04
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Myocardial Ischemia
Keywords: troponin T; CK-MB; protein S-100; Cardiopulmonary Bypass; Erythropoietin
MeSH Terms: conditions — Myocardial Ischemia | interventions — epoetin beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): epoetin beta
  Interventions: Drug: epoetin beta
- 2 (Placebo Comparator): placebo of NaCl
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: epoetin beta — 800UI/kg in 60ml of Nacl IV slow 1 to 3 hours before surgery
  Arms: 1
Drug: placebo — 60ml of NaCl IV slow
  Arms: 2

SUMMARY:
The main objective is to observe the effects of erythropoietin administration on different blood markers of ischaemic cardiac lesions induced by cardiopulmonary bypass.

DETAILED DESCRIPTION:
A new property of erythropoietin (EPO), independent of its hematopoietic role, has recently been discovered. Indeed, it has been reported that this hormone, following binding to its cardiac or cerebral receptors, is able to induce a spectacular cellular protection against ischemic injury. These cardioprotective and neuroprotective effects have been observed experimentally in rodents as well as clinically in humans. In particular, our team has demonstrated that the administration of NeoRecormon® protects the heart against ischemia in the rat by significantly improving its recovery.

In view of these exciting experimental results and of the growing interest of the scientific community for cytoprotective effects of EPO, we are planning the first clinical study examining the cardiac and cerebral protective effects of EPO (NeoRecormon®) in the setting of cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Coronary bypass surgery.
* Surgery not urgent.
* Left ventricular ejection fraction (LVEF) > 40.
* Informed consent form signed.

Exclusion Criteria:

* Valvular surgery.
* Surgery with beating heart, with or without cardiopulmonary bypass.
* Carotid bypass surgery.
* Myocardial infarction less than 30 days.
* Previous history of cardiac surgery.
* Kidney failure (creatinine > 200 µmol/l).
* Uncontrolled hypertension.
* Unstable angina.
* Risk of deep venous thrombosis.
* Vascular cerebral attack less than 30 days.
* Malignant tumour.
* Phenylketonuria.
* Allergy to erythropoietin.
* Previous programmed blood donation.
* Pregnancy and feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Area under curve and maximal plasmatic level of troponin-T, NT-pro-BNP, and creatine kinase-MB (CK-MB) after cardiopulmonary bypass | at anaesthesia (ti), at the end of the cardiopulmonary bypass (t0), puis 6 h, 12 h, 24 h et 48h after the end of the cardiopulmonary bypass

SECONDARY OUTCOMES:
Area under curve and maximal plasmatic level of protein S-100 after cardiopulmonary bypass | at anaesthesia (ti), at the end of the cardiopulmonary bypass (t0), puis 6 h, 12 h, 24 h et 48h after the end of the cardiopulmonary bypass
Blood level of erythropoietin | at injection and 6 hours after the end of cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHAVANON, Pr, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Cardiac Surgery Department - CHU de Grenoble, Grenoble, France

REFERENCES:
- [Background] Bogoyevitch MA. An update on the cardiac effects of erythropoietin cardioprotection by erythropoietin and the lessons learnt from studies in neuroprotection. Cardiovasc Res. 2004 Aug 1;63(2):208-16. doi: 10.1016/j.cardiores.2004.03.017. PMID 15249178
- [Background] Ehrenreich H, Hasselblatt M, Dembowski C, Cepek L, Lewczuk P, Stiefel M, Rustenbeck HH, Breiter N, Jacob S, Knerlich F, Bohn M, Poser W, Ruther E, Kochen M, Gefeller O, Gleiter C, Wessel TC, De Ryck M, Itri L, Prange H, Cerami A, Brines M, Siren AL. Erythropoietin therapy for acute stroke is both safe and beneficial. Mol Med. 2002 Aug;8(8):495-505. PMID 12435860
- [Background] Johnsson P, Backstrom M, Bergh C, Jonsson H, Luhrs C, Alling C. Increased S100B in blood after cardiac surgery is a powerful predictor of late mortality. Ann Thorac Surg. 2003 Jan;75(1):162-8. doi: 10.1016/s0003-4975(02)04318-7. PMID 12537211
- [Background] Joyeux-Faure M, Godin-Ribuot D, Ribuot C. Erythropoietin and myocardial protection: what's new? Fundam Clin Pharmacol. 2005 Aug;19(4):439-46. doi: 10.1111/j.1472-8206.2005.00347.x. PMID 16011730
- [Background] Kerbaul F, Giorgi R, Oddoze C, Collart F, Guidon C, Lejeune PJ, Villacorta J, Gouin F. High concentrations of N-BNP are related to non-infectious severe SIRS associated with cardiovascular dysfunction occurring after off-pump coronary artery surgery. Br J Anaesth. 2004 Nov;93(5):639-44. doi: 10.1093/bja/aeh246. Epub 2004 Sep 3. PMID 15347604